CLINICAL TRIAL: NCT01832571
Title: Open Label Prospective Study of Strategies to Combine Pre-Exposure Prophylaxis (PrEP)With Prevention Efforts
Brief Title: SCOPE: Strategies to Combine PrEP With Prevention Efforts
Acronym: SCOPE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is closed early due to withdrawal of funding. No study procedures were implemented.
Sponsor: FHI 360 (Other)
Collaborators: Family Health Options Kenya (Unknown); Gilead Sciences (Industry); Institute of Tropical Medicine (Other Government); Sex Workers Outreach Programme (Unknown); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 391449
Record Dates: First submitted 2013-04-03; First posted 2013-04-16 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: HIV
Keywords: HIV; PrEP; Female Sex Workers; Kenya
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Once daily Truvada® (Experimental): One tablet of Truvada (200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate) daily
  Interventions: Drug: Once daily Truvada®

INTERVENTIONS:
Drug: Once daily Truvada® — At the enrollment visit, participant's eligibility is assessed per protocol and she is provided with a 30 day supply of Truvada and instructed to take one tablet orally once daily with or without food. Each tablet contains 200 mg emtricitabine (FTC) and 300 mg tenofovir disoproxil fumarate (TDF). Participants will receive Truvada at each clinic visit after it is confirmed that she is HIV negative. There will be a 1 month follow-up visit after enrollment. Thereafter, participants will have quarterly visits until April 2014.
  Other Names: Truvada®

SUMMARY:
This pilot, open-label, prospective study will determine the feasibility of integrating pre-exposure prophylaxis (PrEP) into existing HIV prevention programs for female sex workers and if women who are enrolled in those programs will adhere to the daily PrEP regimen of Truvada®. This study will enroll 500 HIV antibody negative female sex workers in Eldoret and Nairobi, Kenya.

DETAILED DESCRIPTION:
Participants will undergo the following procedures: blood draw for HIV (screening, enrollment, month 1, quarterly follow-up visits and final) and creatinine testing (screening, month 3 and final) and urine pregnancy test (at screening, enrollment and final). At screening, participants will have an HBV antigen test. Information on demographics, sexual behaviors, risk perceptions, partners' HIV status, medical history, PrEP and program acceptability, self-reported adherence to PrEP, alcohol and drug use, depression, social support, stigma, self-efficacy, gender-based violence, contraceptive use, adverse events, and symptoms of potential acute HIV infection will be collected during the study. Detailed information on Truvada for PrEP will be given to the participant and the the participant will be counseled on HIV-risk reduction (according to existing program) during the screening visit. Patient-centered and integrated counseling on HIV risk reduction and PrEP adherence will be conducted at enrollment and follow-up visits. Sexually transmitted infections (STI)will be assessed and treated during visits per local clinical procedures. If a pelvic exam is done per routine clinic procedures, a vaginal and/or endocervical swab will be collected and stored for future research related to HIV infection.

A cohort of 25 systematically-selected participants at each site will have three rounds of in-depth interviews (IDI) to explore the context surrounding many of the study's endpoints. The first IDI will be conducted at the month 1 visit after PrEP initiation. The second IDI will be conducted at the month 3 visit. The third IDI will be conducted at the final study visit.

An IDI will be conducted with all participants at each site who were assigned and willing to use the electronic pill monitoring device (n=25 per site). The purpose of the IDIs is to explore the reasons underlying PrEP use patterns (e.g. the number of times the pill bottle was opened over a specific period of time -- limited, intermittent, or high number of openings). Two rounds of IDIs will be conducted with these participants. The first IDI will be conducted at the month 3 visit and the second at the month 6 visit.

Exit interviews will be conducted with up to 30 participants at each site. Participants may be purposefully selected based on their drug level adherence data or electronic pill measurement data (e.g. low, intermittent, or high PrEP users) or based on other specific issues that emerged over the course of the study (e.g., limited partner support).

Two brief face-to-face (FTF) structured surveys will be administered to all HIV prevention program staff to assess the variables/domains related to the feasibility measures. The first survey will be administered around the initiation of the study and the second survey towards the end of the study. Two interviews will be conducted using a questionnaire with both open- and closed-ended questions, with all counselors and providers, such as nurses, medical officers, and doctors, to gather more in-depth data on the feasibility measures. The first interview will be conducted approximately one month after the first participant is screened and the second interview toward the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willing and able (i.e., successfully complete an open-ended comprehension assessment on key topics related to the study) to give written informed consent
* Expresses willingness at screening and enrollment to take PrEP daily
* Willing to provide contact information and be contacted by staff between visits (per participant-approved methods)
* Is sexually active, defined as having had at least one vaginal sex act in the last four weeks, and reports receiving money or goods in exchange for sex in the last 6 months as part of her source of income/livelihood
* Is HIV antibody negative on rapid test algorithm at the enrollment visit
* Does not have symptoms suggestive of acute HIV infection at the enrollment visit (i.e., fever (temperature above 38ºC), fatigue, sweating, night sweats, pain, rash, pharyngitis, headache, muscle and joint pain, adenopathy (cervical and inguinal), vomiting, diarrhea and coughing) combined with self-reported possibility of recent HIV exposure leading to clinical suspicion of acute HIV infection
* Has a negative urine pregnancy test at screening and enrollment
* Is not currently trying to become pregnant
* Is not breastfeeding
* Has a creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula) at screening
* Is Hepatitis B virus antigen (HBV Ag) negative at screening
* Is in general good health and does not have a medical or social condition which may make study participation unsafe or complicate data interpretation in the opinion of the site investigator
* Is not participating in another PrEP program or PrEP research study
* Is not taking HIV post-exposure prophylaxis at enrollment

Exclusion Criteria:

Pregnant HIV antibody positive Using HIV post-exposure prophylaxis at enrollment

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Drug Adherence | 11 months
  Describe the patterns of adherence to a regimen of daily oral Truvada® among female sex workers currently or newly enrolled in established HIV prevention programs
PrEP Integration | 11 months
  Assess the feasibility of integrating PrEP into existing HIV prevention programs for female sex workers

SECONDARY OUTCOMES:
Assess adherence | 11 months
  Describe self-reported and electronically-monitored patterns of adherence to a regimen of daily oral Truvada® among female sex workers currently or newly enrolled in established HIV prevention programs
drug level adherence | 11 months
  Assess the correlation between drug level adherence data and participant self-reported adherence data
risk-taking behavior | 11 months
  Assess the impact of PrEP on HIV risk-taking behavior
factors affecting Adherence | 11 months
  Identify factors associated with adherence to PrEP
Support of prEP Adherence | 11 months
  Assess impact of adherence support by peer educators on PrEP adherence
Contraceptive Use | 11 months
  Describe Contraceptive Use
Resistance among Seroconverters | 11 months
  Assess resistance to TFV or FTC among seroconverters
Birth Outcomes | 11 months
  Assess birth outcomes among women who choose to continue PrEP during pregnancy
Tenofovir Concentrations | 11 months
  9. Describe tenofovir concentrations among women who choose to continue PrEP during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Deese, MPH, Principal Investigator — FHI 360; Amy Corneli, Ph.D., Principal Investigator — FHI 360
Locations (2):
- Kenya (2):
  - Family Health Options Kenya, Eldoret
  - Sex Workers Outreach Programme (SWOP), Nairobi